CLINICAL TRIAL: NCT02833454
Title: Anterior Cruciate Ligament Reconstruction (ACLR) Using Direct Insertion Technique or Traditional Technique With Single and Double Bundle Procedure.
Brief Title: Study of the Anatomical Direct Insertion Anterior Cruciate Ligament Reconstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Jia-kuo yu, Professor, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DACL-1
Record Dates: First submitted 2016-07-11; First posted 2016-07-14 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2016-07

CONDITIONS: Rupture of Anterior Cruciate Ligament
Keywords: Anterior Cruciate Ligament Reconstruction; Direct Insertion of Anterior Cruciate Ligament
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- direct insertion single bundle ACLR (Active Comparator): Patients with ACL rupture undergo direct insertion anterior cruciate ligament reconstruction using single bundle technique.
  Interventions: Procedure: direct insertion anterior cruciate ligament reconstruction; Procedure: single bundle anterior cruciate ligament reconstruction
- anatomical double bundle ACLR (Experimental): Patients with ACL rupture undergo double bundle anterior cruciate ligament reconstruction.
  Interventions: Procedure: double bundle anterior cruciate ligament reconstruction
- anatomical single bundle ACLR (Experimental): Patients with ACL rupture undergo single bundle anterior cruciate ligament reconstruction.
  Interventions: Procedure: single bundle anterior cruciate ligament reconstruction
- direct insertion double bundle ACLR (Active Comparator): Patients with ACL rupture undergo direct insertion anterior cruciate ligament reconstruction using double bundle technique.
  Interventions: Procedure: direct insertion anterior cruciate ligament reconstruction; Procedure: double bundle anterior cruciate ligament reconstruction

INTERVENTIONS:
Procedure: direct insertion anterior cruciate ligament reconstruction — ACL reconstruction based on direct insertion of ACL.
  Arms: direct insertion double bundle ACLR; direct insertion single bundle ACLR
Procedure: single bundle anterior cruciate ligament reconstruction — anterior cruciate ligament reconstruction using single bundle technique
  Arms: anatomical single bundle ACLR; direct insertion single bundle ACLR
Procedure: double bundle anterior cruciate ligament reconstruction — anterior cruciate ligament reconstruction using double bundle technique
  Arms: anatomical double bundle ACLR; direct insertion double bundle ACLR

SUMMARY:
The purpose of the study is to study the effect of anatomical direct insertion ACL reconstruction compared with conventional anatomical ACL reconstruction.

DETAILED DESCRIPTION:
The investigators divide 320 patients with ACL rupture into 4 groups, each group has 80 patients. The operation technique is different among the groups: group A: conventional anatomical double bundle acl reconstruction, group B: conventional anatomical single bundle acl reconstruction, group DA: direct insertion double bundle acl reconstruction, group DSB: direct insertion single bundle acl reconstruction. The investigators compare the results of the patients of each group at 2 years of surgery.

ELIGIBILITY:
Inclusion Criteria:

* ACL rupture patients aged between 16 to 40 years

Exclusion Criteria:

* combined severe injuries to the operated knee (additional ligament rupture, major meniscus loss, patella instability, cartilage damage >2°, pathologic leg axis deviation)
* any injury or surgery to the contralateral knee
* any infammatory or systemic disease, neuromuscular disease in the lower limbs, any recent knee infection

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 320 (Estimated)
Dates: Start 2016-07; Primary Completion 2018-07 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Lysholm score of the knee | two years
  Lysholm score of the knee was evaluated preoperatively and at 2 years post operation .
  Scale name:score
Tegner score of the knee | two years
  Tegner score of the knee was evaluated preoperatively and at 2 years post operation .
  Scale name:score
IKDC score of the knee | two years
  IKDC score of the knee was evaluated preoperatively and at 2 years post operation .
  Scale name:score

SECONDARY OUTCOMES:
KT-2000 of the knee | two years
  KT-2000 of the knee was evaluated preoperatively and at 2 years post operation.

CONTACTS AND LOCATIONS:
Overall Officials: Jia-Kuo Yu, MD, Study Chair — Peking University Third Hospital